CLINICAL TRIAL: NCT07199270
Title: A Randomized, Double-blind, Placebo-controlled of GR2303 Injection in Healthy Adult Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Pharmacologic of GR2303
Brief Title: A Study to Evaluate the Safety, Immunogenicity, and Pharmacokinetics of GR2303 in Healthy Adult
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR2303-001
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Health Adult Subjects
Keywords: Inflamatory bowel disease; phase 1; GR2303

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- group 1 (Experimental): single dose
  Interventions: Biological: GR2303 injection; Biological: Placebo
- group 2 (Experimental): single dose
  Interventions: Biological: GR2303 injection; Biological: Placebo
- group 3 (Experimental): single dose
  Interventions: Biological: GR2303 injection; Biological: Placebo
- group 4 (Experimental): single dose
  Interventions: Biological: GR2303 injection; Biological: Placebo
- group 5 (Experimental): single dose
  Interventions: Biological: GR2303 injection; Biological: Placebo
- group 6 (Experimental): multiple dose
  Interventions: Biological: GR2303 injection; Biological: Placebo
- group 7 (Experimental): multiple dose
  Interventions: Biological: GR2303 injection; Biological: Placebo
- group 8 (Experimental): multiple dose
  Interventions: Biological: GR2303 injection; Biological: Placebo

INTERVENTIONS:
Biological: GR2303 injection — single dose
  Arms: group 1; group 2; group 3; group 4; group 5
Biological: Placebo — single dose
  Arms: group 1; group 2; group 3; group 4; group 5
Biological: GR2303 injection — multiple dose
  Arms: group 6; group 7; group 8
Biological: Placebo — multiple dose
  Arms: group 6; group 7; group 8

SUMMARY:
he goal this clinical trail is to evaluate the safety、Pharmacokinetic and immunogenicity of GR2303 injection。 Subjects will be enrolled in different groups in sequential order, and within each group will be randomly assigned to receive either GR2303 injection or placebo administration, with each Subjects will be enrolled in only one of these groups

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics, and preliminary pharmacodynamic profile of GR2303 Injection in healthy adult Chinese subjects.

After signing the informed consent form, subjects who meet the criteria for enrollment will be entered into different groups according to the randomization number. Subjects will be enrolled in only one of these groups.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects
2. Signed informed consent

Exclusion Criteria:

1. History or presence of any clinically significant organ system disease that could interfere with the objectives of the study or the safety of the subjects.
2. Prior use of drug targeting TNF-like cytokine 1A
3. history of malignant tumor
4. psitive results for Hepatitis B surface antigen (HBsAg), anti Hepatitis C antibody (HCV Ab) or human immunodeficiency virus (HIV)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 16 weeks

SECONDARY OUTCOMES:
Cmax | 16 weeks
Tmax | 16 weeks
t 1/2 | 16 weeks
ADA | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No